CLINICAL TRIAL: NCT01940133
Title: Phase I Study of Oral PQR309 in Patients With Advanced Solid Tumors
Brief Title: A Study to Investigate Safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) of PQR309
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PIQUR Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQR309-001; 2013-003441-42 (EudraCT Number)
Record Dates: First submitted 2013-09-06; First posted 2013-09-12 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PQR309 (Experimental): Different dose evaluation
  Interventions: Drug: PQR309

INTERVENTIONS:
Drug: PQR309 — Dosing will be orally, once a day for the duration of the trial.

SUMMARY:
This study is a Phase I, open label study to determine the Maximum Tolerated Dose(MTD) and the Recommended Phase II Dose (RP2D) in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumor for which no therapy of proven efficacy is available.
* Age ≥ 18
* Evidence of tumor progression with measurable or evaluable disease.
* Use of adequate contraceptive measures for male patients.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1.
* Signed informed consent.

Exclusion Criteria:

* Concomitant anticancer therapy (e.g., chemotherapy, radiotherapy, hormonal, immunotherapy, biological response modifier, signal transduction inhibitors)
* Patients with a history of myocardial infarction or coronary artery bypass within the last 3 years.
* Patients with severe/unstable angina, coronary/peripheral arterial bypass, symptomatic congestive heart failure NYHA Class 3 or 4, hypertension BP>150/100mmHg.
* Pre-diagnosed diabetes mellitus.
* Fasting glucose > 7.0 mmol/L or HbA1c > 6%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and the Recommended Phase II Dose (RP2D) | In average 1 year

SECONDARY OUTCOMES:
To determine overall safety | 1 year
  Incidence of SAEs, incidence and severity of all AEs, changes of vital signs, physical examinations, body weight, changes of routine laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Wicki, Dr., Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Wicki A, Brown N, Xyrafas A, Bize V, Hawle H, Berardi S, Cmiljanovic N, Cmiljanovic V, Stumm M, Dimitrijevic S, Herrmann R, Pretre V, Ritschard R, Tzankov A, Hess V, Childs A, Hierro C, Rodon J, Hess D, Joerger M, von Moos R, Sessa C, Kristeleit R. First-in human, phase 1, dose-escalation pharmacokinetic and pharmacodynamic study of the oral dual PI3K and mTORC1/2 inhibitor PQR309 in patients with advanced solid tumors (SAKK 67/13). Eur J Cancer. 2018 Jun;96:6-16. doi: 10.1016/j.ejca.2018.03.012. Epub 2018 Apr 13. PMID 29660598